CLINICAL TRIAL: NCT00135395
Title: A Phase IIIb, Open -Label, Randomized Multi-center Study Comparing the Antiviral Efficacy, Safety, and Effect on Serum Lipids of Atazanavir/Ritonavir Versus Lopinavir/Ritonavir, in Combination With Two Nucleoside or Nucleotide Reverse Transcriptase Inhibitors (NRTIs) in HIV-1 Infected Subjects Experiencing Their First Virologic Failure While Receiving a NNRTI-containing HAART Regimen.
Brief Title: A Phase IIIb Study Comparing Two Boosted Protease Inhibitor-based HAART Regimens in HIV-infected Patients Experiencing Their First Virologic Failure While Receiving an NNRTI-containing HAART Regimen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI424-103
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2008-07

CONDITIONS: HIV Infections
Keywords: HIV/AIDS; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — atazanavir, ritonavir drug combination; Atazanavir Sulfate; Lopinavir

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Atazanavir+ritonavir
- B (Active Comparator)
  Interventions: Drug: Lopinavir+ritonavir

INTERVENTIONS:
Drug: Atazanavir+ritonavir — Capsules, Oral, 300mg/100mg, once daily, 24 weeks.
  Other Names: Reyataz
  Arms: A
Drug: Lopinavir+ritonavir — Capsules, Oral, 800mg/200mg, twice daily, 24 weeks.
  Arms: B

SUMMARY:
The purpose of this study is to compare the anti-HIV efficacy, safety and effect of serum lipids of two boosted protease inhibitor-based HAART regimens (ARV/RTV v. LPV/RTV) in HIV-1 infected subjects who have experienced their first virologic failure while receiving a NNRTI-containing HAART regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age infected with HIV
* Plasma HIV RNA ≥ 1000 copies/mL and CD4 cell count ≥ 50 cells/mm3
* Currently receiving a NNRTI-containing HAART regimen or not currently receiving a NNRTI-containing HAART regimen and have not been treated with an alternative regimen since the documented virologic failure (with genotype performed within 2 weeks of the discontinuation of the failing regimen and the genotype report is available)
* The failing NNRTI-containing regimen must be the patient's first virologic failure on treatment and contain a NNRTI and at least 2 NRTIs. The regimen must have been administered for at least 24 weeks and the patient must have documented virologic response to the regimen (HIV RNA < 400 c/mL)

Exclusion Criteria:

* Pregnancy or breastfeeding
* Reported virologic failure to two or more antiretroviral regimens
* Active AIDS-defined opportunistic infection or disease
* Proven or suspected acute hepatitis within 30 days prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2004-05; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Co-Primary Outcomes in this study 1)Viral load reduction from baseline through Week 24 2)Change in lipids from baseline at Week 12

SECONDARY OUTCOMES:
Viral load reduction from baseline at Weeks 48,72,96;Subjects with HIV RNA<50 and <400 c/mL at Weeks 24,48,72 & 96;Patterns of resistance;Safety and tolerability through Week 96 including fasting lipid values;Adherence at Weeks 4,12,24,48,72 & 96.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (53):
- United States (52):
  - Local Institution, Hobson City, Alabama
  - Local Institution, Montgomery, Alabama
  - Local Institution, Phoenix, Arizona
  - Local Institution, Little Rock, Arkansas
  - Local Institution, Bakersfield, California
  - Local Institution, Los Angeles, California
  - Local Institution, San Francisco, California
  - Local Institution, San Mateo, California
  - Local Institution, Tarzana, California
  - Local Institution, West Hollywood, California
  - Local Institution, Norwalk, Connecticut
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Atlantis, Florida
  - Local Institution, Fort Lauderdale, Florida
  - Local Institution, Jacksonville, Florida
  - Local Institution, Miami, Florida
  - Local Institution, Miami Beach, Florida
  - Local Institution, North Miami, Florida
  - Local Institution, Orlando, Florida
  - Local Institution, Plantation, Florida
  - Local Institution, Safety Harbor, Florida
  - Local Institution, Tampa, Florida
  - Local Institution, Atlanta, Georgia
  - Local Institution, Decatur, Georgia
  - Local Institution, Chicago, Illinois
  - Local Institution, Indianapolis, Indiana
  - Local Institution, Louisville, Kentucky
  - Local Institution, New Orleans, Louisiana
  - Local Institution, Boston, Massachusetts
  - Local Institution, Springfield, Massachusetts
  - Local Institution, Berkley, Michigan
  - Local Institution, Jackson, Mississippi
  - Local Institution, St Louis, Missouri
  - Local Institution, Las Vegas, Nevada
  - Local Institution, East Orange, New Jersey
  - Local Institution, Hillsborough, New Jersey
  - Local Institution, Jersey City, New Jersey
  - Local Institution, Brooklyn, New York
  - Local Institution, Mount Vernon, New York
  - Local Institution, New York, New York
  - Local Institution, Valhalla, New York
  - Local Institution, Greenville, North Carolina
  - Local Institution, Huntersville, North Carolina
  - Local Institution, Winston-Salem, North Carolina
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Columbia, South Carolina
  - Local Institution, Dallas, Texas
  - Local Institution, Galveston, Texas
  - Local Institution, Harlingen, Texas
  - Local Institution, Houston, Texas
  - Local Institution, Hampton, Virginia
- Local Institution, Santruce, Puerto Rico